CLINICAL TRIAL: NCT01760681
Title: A Randomized Sham-Controlled Study of H-Coil Repetitive Transcranial Magnetic Stimulation for Treatment-Resistant Late-Life Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHA-14-12
Record Dates: First submitted 2012-12-18; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2012-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- H coil DTMS (Experimental): 20 daily deep TMS treatments
  Interventions: Device: H- Coil DTMS
- inactive stimulation (Sham Comparator): 20 daily sham deep TMS treatments
  Interventions: Device: Sham

INTERVENTIONS:
Device: H- Coil DTMS — 20 daily deep rTMS treatments
  Other Names: H1 coil DTMS
  Arms: H coil DTMS
Device: Sham
  Other Names: inactive treatment
  Arms: inactive stimulation

SUMMARY:
The purpose of the study is to explore the efficacy and safety of H-Coil rTMS in comparison to a sham H-Coil rTMS in older patients with treatment-resistant major depressive disorder.Subjects will be randomized to receive H1-Coil rTMS or sham H1-Coil rTMS. The acute treatment phase will last four weeks. Treatment is administered daily, 5 days per week (i.e., 20 treatments). Depressive symptoms will be assessed using the HDRS-24. If subjects achieve the pre-defined primary outcome criteria of remission (HDRS-24 score < 10 and 60% reduction in symptoms) they will continue with twice weekly treatment for two more weeks to ensure the durability of the remission. Subjects who do not achieve remission will exit the study after the acute treatment phase of four weeks. The blind will not be broken to subjects until the completion of the study

ELIGIBILITY:
Inclusion Criteria:

1. are outpatients
2. are voluntary and competent to consent to treatment
3. have a Structured Clinical Interview for DSM-IV (SCID)103 confirmedn DSM-IV diagnosis of MDD, single or recurrent
4. are between the ages of 60 and 85
5. have failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of > 3 in the current episode 104, 105 OR have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF 1 or 2)
6. have a score > 22 on the HDRS-24
7. have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening
8. able to adhere to the treatment schedule
9. Pass the TMS safety screening questionnaire
10. have normal thyroid functioning based on pre-study blood work.

Exclusion Criteria:

1. have a history of DSM-IV substance dependence or abuse within the last 3 months
2. have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
3. are acutely suicidal
4. are pregnant
5. have a lifetime SCID diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms
6. have a SCID diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder) assessed by a study investigator to be primary and causing greater impairment than MDD
7. have a SCID diagnosis of any personality disorder and assessed by a study investigator to be primary and causing greater impairment than MDD
8. have presumed or probable dementia, as defined by Mini Mental Status Exam (MMSE) < 26 and clinical evidence of dementia. Patients screened out due to possible dementia will be referred to the local memory clinic for evaluation to clarify the presence or absence of dementia
9. have failed a course of ECT within the current depressive episode
10. have received rTMS for any previous indication due to the potential compromise of subject blinding
11. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes
12. on a dose of Buproprion greater than 300mg per day
13. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
14. if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
15. clinically significant laboratory abnormality, in the opinion of the investigator
16. currently (or in the last 4 weeks) take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy
17. inability to communicate
18. non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in depression symptoms, evaluated by HDRS | 6-8 weeks
  Clinical antidepressant response at the end of the treatment, define as a decline in Hamilton depression rating scale (HDRS-24) from the baseline rating by 50%.

SECONDARY OUTCOMES:
1. Remission in depression | 6-8 weeks
  1. Clinical antidepressant remission at the end of the treatment, define as exit HDRS-24 <10 and 60% reduction in total score.

CONTACTS AND LOCATIONS:
Locations (1):
- shalvataMHC, Hod HaSharon, Israel